CLINICAL TRIAL: NCT04550403
Title: Clinical Phenotype and Outcomes of Inpatients With COVID-19 and Diabetes
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Riccardo Bonadonna, Head of Endocrinology and metabolic diseases unit, Azienda Ospedaliero-Universitaria di Parma
Other Study IDs: 27557
Record Dates: First submitted 2020-09-10; First posted 2020-09-16 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus; Covid19
Keywords: diabetes; Covid-19; inhospital mortality; intensive care unit
MeSH Terms: conditions — Diabetes Mellitus; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with diabetes have been listed as people at higher risk for severe illness from COVID-19. Moreover, the relationship between diabetes-related phenotypes and the severity of COVID-19 remains unknown. This observational study aims to to evaluate the risk of disease severity and mortality in association with diabetes in COVID-19 inpatients and identify the clinical and biological features associated with worse outcomes.

DETAILED DESCRIPTION:
The epidemic of coronavirus disease-2019 (COVID-19), a disease caused by the severe acute respiratory syndrome-coronavirus-2 (SARS-CoV-2) virus, rapidly spread worldwide and was declared a pandemic by the World Health Organization on 11 March 2020.

It is well known that people with diabetes have increased infection risk, especially for influenza and pneumonia. Moreover, diabetes was previously reported as a major risk factor for mortality in people infected with the H1N1 pandemic influenza and, more recently, with the Middle East respiratory syndrome-related coronavirus (MERS-CoV) . Epidemiological studies have quickly and consistently pointed out diabetes as one of the major comorbidities associated with COVID-19 and affecting its severity.

The prevalence of diabetes in patients with COVID-19 was first reported to range from 5% to 20%. Furthermore, the COVID-19-Associated Hospitalisation Surveillance Network (COVID-NET) reported a diabetes prevalence of 28.3% in hospitalised patients in the USA.

More importantly, all studies published so far have reported a two- to threefold higher prevalence of diabetes in patients in ICUs compared with those with less severe disease and an increased mortality in people with diabetes. A recent meta-analysis further demonstrated that diabetes was associated with a more than doubled risk for ICU admission and a more than tripled risk for death.

However, precise data regarding diabetes characteristics in hospitalised people with COVID-19 are still lacking. Moreover, the relationship between diabetes-related phenotypes and the severity of COVID-19 remains unknown. This study aims to identify the clinical and biological features and potential interactions of diabetic therapies associated with disease severity and mortality risk in people hospitalised for COVID-19. Hospital medical records of inpatients, hospitalized between February 23 to March 31 2020, at the Internal Medicine Unit dedicated to COVID-19 in the Academic Hospital of Parma, Italy will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* admission with COVID-19 to the Internal Medicine Unit dedicated to COVID-19 (Macrounit 1), academic hospital in Parma (Italy) between February 23 to March 31 2020.

Exclusion Criteria:

* during hospitalization inter or intra-hospital transfer of inpatients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with and without diabetes, hospitalized for COVID-19 between February 23 to March 31 2020, at the Internal Medicine Unit dedicated to COVID-19 in the Academic Hospital of Parma, Italy
Sampling Method: Probability Sample
Enrollment: 757 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
prevalence of intensive care unit admission and/or in-hospital mortality among COVID-19 inpatients | february 23 to march 31, 2020
  to assess risk of intensive care unit admission and/or death among COVID-19 inpatients

SECONDARY OUTCOMES:
prevalence of death among COVID-19 inpatients with and without diabetes | february 23 to march 31, 2020
  to compare risk of death among inpatients in presence or absence of diabetes
prevalence of intensive care unit admission among COVID-19 inpatients with and without diabetes | february 23 to march 31, 2020
  to compare intensive care unit admission among inpatients in presence or absence of diabetes
demographic and clinical characteristics (age,gender, comorbidity status) and death and/or intensive care unit admission during hospitalization | february 23 to march 31, 2020
  to identify socio-demographic as predictors of severe prognosis (death or intensive care unit admission) during hospitalization
laboratory parameters (glycated hemoglobin, glucose at admission, renal and liver function markers, blood count, inflammatory markers, hemostasis) and death and/or intensive care unit admission during hospitalization | february 23 to march 31, 2020
  to identify laboratory variables as predictors of severe prognosis (death or intensive care unit admission) during hospitalization
pharmacological therapies and death and/or intensive care unit admission during hospitalization | february 23 to march 31, 2020
  to identify pharmacological therapies as predictors of severe prognosis (death or intensive care unit admission) during hospitalization
number of days of hospitalization in patients with and without diabetes | february 23 to march 31, 2020
  to compare total length of hospitalization in patients with or without diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Bonadonna, MD, PhD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma
Locations (1):
- Endocrinology and metabolic diseases Unit, Parma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Memish ZA, Perlman S, Van Kerkhove MD, Zumla A. Middle East respiratory syndrome. Lancet. 2020 Mar 28;395(10229):1063-1077. doi: 10.1016/S0140-6736(19)33221-0. Epub 2020 Mar 4. PMID 32145185
- [Background] Bindom SM, Lazartigues E. The sweeter side of ACE2: physiological evidence for a role in diabetes. Mol Cell Endocrinol. 2009 Apr 29;302(2):193-202. doi: 10.1016/j.mce.2008.09.020. Epub 2008 Oct 1. PMID 18948167
- [Background] Yang JK, Lin SS, Ji XJ, Guo LM. Binding of SARS coronavirus to its receptor damages islets and causes acute diabetes. Acta Diabetol. 2010 Sep;47(3):193-9. doi: 10.1007/s00592-009-0109-4. Epub 2009 Mar 31. PMID 19333547
- [Background] Drucker DJ. Coronavirus Infections and Type 2 Diabetes-Shared Pathways with Therapeutic Implications. Endocr Rev. 2020 Jun 1;41(3):bnaa011. doi: 10.1210/endrev/bnaa011. PMID 32294179
- [Background] Wang B, Li R, Lu Z, Huang Y. Does comorbidity increase the risk of patients with COVID-19: evidence from meta-analysis. Aging (Albany NY). 2020 Apr 8;12(7):6049-6057. doi: 10.18632/aging.103000. Epub 2020 Apr 8. PMID 32267833